CLINICAL TRIAL: NCT05883410
Title: The Effect of Proprioceptive Neuromuscular Facilitation-Based Stretching and Mulligan Mobilization on Kinesiophobia and Proprioception in Wrist Joint Limitation After Distal Radius End Fractures
Brief Title: The Effect of Two Different Protocol in Wrist Joint Limitation After Distal Radius End Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Zeynep HOŞBAY, Associate Professor, Physiotherapist, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Biruni Uni
Record Dates: First submitted 2023-04-13; First posted 2023-06-01 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Distal Radius Fracture; Wrist Fracture
Keywords: Distal Radius Fractures; Joint Limitation; Mulligan Mobilization; PNF Technique; Proprioception
MeSH Terms: conditions — Wrist Fractures | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Who Masked: Participant
Masking Description: Participants does not know which type of treatment is received themselves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF Treatment Group (Experimental): Hold-relax is a PNF technique will be applied to this group.
  Interventions: Other: Exercise; Other: PNF Technique
- Mulligan Mobilization Treatment (Active Comparator): The Mobilization with movement (MWM) technique will be applied to this group.
  Interventions: Other: Exercise; Other: Mulligan Mobilization

INTERVENTIONS:
Other: Exercise — It is important for the therapist to organize a home exercise program to provide edema and pain control. The exercise program should be specific and clear to the patient. The exercise program will be taught to the patient and given as a home program
  Other Names: Traditional Exercise Program
Other: PNF Technique — While the limb is in the agonist pattern, the patient is instructed to perform isometric contractions for 5-8 seconds against maximum resistance without movement at the limiting point. After maximum isometric contraction, the patient is instructed to actively relax.Participants in the second group will be applied 10 repetitions of isometric contractions for 8 seconds at the limitation points of the movement with the PNF techniques, the hold and relax active movement technique in the direction of wrist flexion and extension.
  Arms: PNF Treatment Group
Other: Mulligan Mobilization — In thw Mobilization with movement technique; the patient is expected to perform painless ROM. After obtaining painless movement in the patients participating in the study, this application will be applied to the patient with the painless active movement technique in 10 repetitions and 2-3 sets. Rest time between sets will be 15-20 seconds. Patients will be taught self-mobilization to ensure the continuity of painless movement. Self-mobilization will be applied by the patient at home with 10 repetitions every two hours (29).
  Arms: Mulligan Mobilization Treatment

SUMMARY:
Distal radius fractures are among the most common fractures treated by hand therapists. These patients are most conservatively treated with closed reduction and cast immobilization. Since there is an immobilization process after both treatments, a limitation in the range of motion of the joint occurs in patients. For this reason, most of the treatment models applied in rehabilitation are about restoring the range of motion of the joint. In general, kinesiophobia occurs due to joint limitation and pain. Loss of proprioception occurs in patients with mobility and desire as a result of kinesiophobia. By investigating the techniques used in rehabilitation, the more correct one for the patient can be selected. There is no clear result in the literature about which of the application methods is more effective. The aim of the study is to compare the effects of proprioceptive neuromuscular facilitation (PNF) based stretching and Mulligan mobilization on pain, proprioception (joint position sense), wrist functionality, muscle strength and kinesiophobia in patients with joint limitation after distal radius end fracture. Thirty-four individuals aged 18-65 who were referred to a physiotherapy and rehabilitation program after distal radius end fracture will be included in the study. Individuals will be randomized into two groups. In the study, algometer and Visual Analogue Scale (VAS) were used to evaluate the pain intensity of the patients, universal goniometer for the evaluation of the forearm and wrist joint range of motion, microFET®2 Digital Handheld Dynamometer for the evaluation of the strength of the wrist flexor and extensor muscles, ulnar and radial deviation muscles. device will be used. The functional use of the wrist of the individuals is using the patient-based wrist assessment questionnaire (Patient Graded Wrist Assessment PRWE), the sense of attachment position for proprioception, and the Tampa Kinesiophobia Scale (TKS) for kinesiophobia. In our study, an exercise program will be applied with a physiotherapist for 6 weeks, 2 days a week, 45 minutes. To the first group; In addition to the traditional treatment, Mulligan mobilization will be applied, and the second group will be applied to the PNF techniques, 'hold-relax' in addition to the traditional treatment. It can be considerable that both techniques applied in our study may have positive effects on pain, kinesiophobia and proprioception.

DETAILED DESCRIPTION:
The wrist has a complex anatomy and consists of the following structures; bone, ligament, musculotendinous and neurovascular. The distal ends of the radius and ulna are radio-ulnar, radio-carpal and ulno-carpal; carpal bones form midcarpal joints among themselves (1).

The ulna and radius bones articulate with the wrist bones on the distal side, thus providing bony integrity (2).

The wrist joint is the joint region that is most exposed to trauma. Radius distal end fractures account for approximately 20% of fractures admitted to the emergency department and 75% of all forearm fractures. (3).

Distal radius fractures are very common, alone or in combination with other fractures and injuries. For example, in the United States there is an incidence of approximately 67 upper extremity fractures per 10,000 persons per year. Distal radius and ulna fractures account for approximately 25% of all fractures (4).

Distal radius fractures can occur at any age, with a largely bimodal distribution based on age and gender; They are children under 18 and adults over 50 (5).

The overall incidence of DR tip fractures occurring each year is increasing worldwide. For example, a 1998 study by Melton et al. of Rochester, Minnesota, USA documented a 17% increase in DR fractures between 1945 and 1994 (6). Direct trauma is less common in distal radius fractures.

It occurs as a result of direct hitting and impact blows to the distal radius (7). Indirect trauma is more common. Individuals consciously or unconsciously position their elbows in extension, their forearms in pronation, and their wrists in dorsiflexion, and this position, which is defined as falling on an open hand, causes fractures (8). It is very important to determine both the type of fracture and the level of injury well. Thus, the treatment will be easier and the healing process will be accelerated (9).

Fracture healing has been studied in different phases by the researchers. As it is generally known, it consists of three phases; Inflammatory phase, Repair phase, Remodeling phase (10-13).

All these processes require prostaglandins and bone stimulants, which are binding factors. (14,15). According to Wolf's law, skeletal mass and strength are variable according to load distribution (16). It has been observed that compressive axial loads stimulate periosteal callus formation. Shearing and tensile forces have been shown to inhibit union (17).

Displacement, deformation and loads at the fracture site affect the behavior of bone cells, tissue structure, and thus healing. (18).

The primary goals of treatment are to control edema and pain, and to restore normal range of motion to the patient (19). Restoring joint play in patients with resistant joint stiffness will be important in gaining joint range of motion (ROM). Joint mobilization techniques can be used for this purpose (20,21). Movement mobilization (MWM) technique unique to Mulligan Concept, which is one of the mobilization techniques, can be applied safely and effectively in both musculoskeletal and nervous system diseases. Mulligan Concept is functional restoration, techniques are applied in functional positions to improve the daily functions of patients (22).

Stretching, which is a frequently applied method for gaining ROM, can be added to the exercise program as long as fracture healing allows, and by obtaining the opinion of the surgeon with the radiographic findings. In the literature, it has been reported that passive stretching lasting 30 seconds has positive effects on ROM gain when performed repeatedly during the day (23). One of the stretching techniques, Proprioceptive Neuromuscular Facilitation (PNF) based stretching, which is based on the neurophysiological mechanisms of reciprocal innervation and post-isometric relaxation, is one of the active stretching applications that improves mobility, movement control and joint coordination. (24,25).

The consequences of traumatic wrist lesions contribute to proprioceptive and motor control deficits observed in both the acute and post-acute period (26). The aim of rehabilitation after distal radius end fracture is to restore joint mobility and functionality, reduce pain and edema, increase muscle activity through active movement, and train proprioception (27)

Adding mobilization and PNF hold-loose technique to the traditional treatment program may be beneficial in terms of pain, proprioception, muscle strength and kinesiophobia after distal radius end fracture, but it is not known which method will improve more in this patient group. (28).

The aim of the study is to compare the effects of proprioceptive neuromuscular facilitation (PNF) based stretching and Mulligan mobilization on pain, proprioception (joint position sense), wrist functionality, muscle strength and kinesiophobia in patients with joint limitation after distal radius end fracture.

ELIGIBILITY:
Inclusion Criteria:

* To be directed to the physiotherapy program after distal radius fracture between the ages of 18-65,
* Having signed the Informed Consent Form
* Patients with good cooperation level

Exclusion Criteria:

* Being illiterate of reading and writing
* Having another orthopedic, neurological and cardiovascular problem
* Pre-existing complex regional pain syndrome
* Having had an operation involving the ipsilateral upper extremity in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Pain Threshold Assessment | 10 minutes
  The pressure pain threshold in the wrist joint will be recorded by measuring with the Baseline Dolorimeter 66 pounds. In addition to subjective assessment methods, it is necessary to record before and after treatment using this device in order to evaluate pain more objectively and to be expressed in the literature as data with high scientific evidence level.
Visual Analog Scale | 10 minutes
  Visual Analog Scale (VAS) can be used to assess pain which perceived by patients. . VAS is a frequently used scale that indicates the severity of pain numerically. A 10 cm line is divided into 10 equal parts and both ends are numbered from 0 to 10 as the least and maximum pain intensity. Patients are asked to mark the place that best suits their pain intensity.
Muscle Strength Assessment | 8 minutes
  It is planned to use microFET®2 Digital Handheld Dynamometer device to evaluate the strength of wrist flexor and extensor muscles, ulnar and radial deviation muscles. The device has the feature of acquiring objective data and transferring it to a computer. Measurements are recorded in the range of 0-300 lbs. Measurements will be tested with 10 seconds of resistance in the muscle test position. The data of this device are needed to express the weakness in the wrist muscles after the distal radius end fracture as a quantitative value. Thus, the effectiveness of treatment programs can be compared by showing the effect of decreasing muscle strength.
Range of Motion Assessment (ROM) | 10 minutes
  The forearm and wrist joint range of motions will be performed with a universal goniometer in the patient sitting position and on the forearm examination table as degree. Evaluation will take place at weeks 6 and 12 (30-33).
Proprioception Assessment | 8 minutes
  The sensation of kinesthesia is measured by perceiving the minimum degree of motion of the joint per unit time and is generally used as the "passive motion detection threshold" in studies. Joint position sense; It is measured by the ability of a joint at a certain angle to actively or passively repeat the same position. As the error made while repeating the determined target angle decreases, the quality of the sense of joint position increases. Goniometer will be used for evaluation. The patients' deviations from the target angles for the wrist will be recorded as degree (33-37).
Tampa Kinesiophobia Scale | 10 minutes
  It will be used to assess kinesiophobia. The Tampa Kinesiophobia Scale is a self-report measure developed to assess the fear of movement-related pain in patients with musculoskeletal pain. Its items are grouped as activity avoidance and somatic focus, according to two different factors (38,39).The scale is scored with range from 1-4, the negatively worded items are 4,8,12,1 and having a reverse scoring (4-1). The 17 item total scores are ranged from 17 to 68 where the lowest 17 means no kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia

SECONDARY OUTCOMES:
Patient Rated Wrist Evaluation (PRWE) | 10 minutes
  It will be used to evaluate the functionality of patients. The Patient Based Wrist Evaluation (PRWE) is a questionnaire used to determine the level of pain and disability in hand/wrist problems. It includes pain and function subsections and specific activities and daily activities sections. It consists of 15 questions and is a subjective evaluation result scale. The validity and reliability of the scale were determined by evaluating distal radius fractures and wrist injuries. Each response is scored from 0 to 10 (0 = no pain/no difficulty; 10 = maximum pain felt/no ability to do anything). The total score is calculated out of 100, and a high score indicates a higher level of disability (40,41).

CONTACTS AND LOCATIONS:
Overall Officials: İrem Guney, PT, Study Chair — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bruder AM, Taylor NF, Dodd KJ, Shields N. Physiotherapy intervention practice patterns used in rehabilitation after distal radial fracture. Physiotherapy. 2013 Sep;99(3):233-40. doi: 10.1016/j.physio.2012.09.003. Epub 2012 Nov 30. PMID 23200599
- [Result] Brown PW. Body and soul. J Hand Ther. 1996 Jul-Sep;9(3):201-2. doi: 10.1016/s0894-1130(96)80082-2. No abstract available. PMID 8856564
- [Result] Chen NC, Jupiter JB. Management of distal radial fractures. J Bone Joint Surg Am. 2007 Sep;89(9):2051-62. doi: 10.2106/JBJS.G.00020. No abstract available. PMID 17768207
- [Result] Karagiannopoulos C, Sitler M, Michlovitz S, Tierney R. A descriptive study on wrist and hand sensori-motor impairment and function following distal radius fracture intervention. J Hand Ther. 2013 Jul-Sep;26(3):204-14; quiz 215. doi: 10.1016/j.jht.2013.03.004. Epub 2013 Apr 28. PMID 23628557
- [Result] Cruess RL, Dumont J. Fracture healing. Can J Surg. 1975 Sep;18(5):403-13. PMID 1175109
- [Result] Frost HM. Mechanical determinants of bone modeling. Metab Bone Dis Relat Res. 1982;4(4):217-29. doi: 10.1016/0221-8747(82)90031-5. PMID 6763662
- [Result] Ilyas AM, Jupiter JB. Distal radius fractures--classification of treatment and indications for surgery. Orthop Clin North Am. 2007 Apr;38(2):167-73, v. doi: 10.1016/j.ocl.2007.01.002. PMID 17560399
- [Result] Jerrhag D, Englund M, Karlsson MK, Rosengren BE. Epidemiology and time trends of distal forearm fractures in adults - a study of 11.2 million person-years in Sweden. BMC Musculoskelet Disord. 2017 Jun 2;18(1):240. doi: 10.1186/s12891-017-1596-z. PMID 28576135
- [Result] Khan SN, Bostrom MP, Lane JM. Bone growth factors. Orthop Clin North Am. 2000 Jul;31(3):375-88. doi: 10.1016/s0030-5898(05)70157-7. PMID 10882464
- [Result] Youdas JW, Krause DA, Egan KS, Therneau TM, Laskowski ER. The effect of static stretching of the calf muscle-tendon unit on active ankle dorsiflexion range of motion. J Orthop Sports Phys Ther. 2003 Jul;33(7):408-17. doi: 10.2519/jospt.2003.33.7.408. PMID 12918866
- [Result] Schier JS, Chan J. Changes in life roles after hand injury. J Hand Ther. 2007 Jan-Mar;20(1):57-68; quiz 69. doi: 10.1197/j.jht.2006.10.005. PMID 17254909
- [Result] Safi A, Hart R, Teknedzjan B, Kozak T. Treatment of extra-articular and simple articular distal radial fractures with intramedullary nail versus volar locking plate. J Hand Surg Eur Vol. 2013 Sep;38(7):774-9. doi: 10.1177/1753193413478715. Epub 2013 Feb 26. PMID 23442339
- [Result] Reyhan AC, Sindel D, Dereli EE. The effects of Mulligan's mobilization with movement technique in patients with lateral epicondylitis. J Back Musculoskelet Rehabil. 2020;33(1):99-107. doi: 10.3233/BMR-181135. PMID 31104005
- [Result] Reid SA, Andersen JM, Vicenzino B. Adding mobilisation with movement to exercise and advice hastens the improvement in range, pain and function after non-operative cast immobilisation for distal radius fracture: a multicentre, randomised trial. J Physiother. 2020 Apr;66(2):105-112. doi: 10.1016/j.jphys.2020.03.010. Epub 2020 Apr 11. PMID 32291223
- [Result] de Palma L, Tulli A, Maccauro G, Sabetta SP, del Torto M. Fracture callus in osteopetrosis. Clin Orthop Relat Res. 1994 Nov;(308):85-9. PMID 7955707
- [Result] Ozaki A, Tsunoda M, Kinoshita S, Saura R. Role of fracture hematoma and periosteum during fracture healing in rats: interaction of fracture hematoma and the periosteum in the initial step of the healing process. J Orthop Sci. 2000;5(1):64-70. doi: 10.1007/s007760050010. PMID 10664441
- [Result] Noordeen MH, Lavy CB, Shergill NS, Tuite JD, Jackson AM. Cyclical micromovement and fracture healing. J Bone Joint Surg Br. 1995 Jul;77(4):645-8. PMID 7615614
- [Result] Melton LJ 3rd, Amadio PC, Crowson CS, O'Fallon WM. Long-term trends in the incidence of distal forearm fractures. Osteoporos Int. 1998;8(4):341-8. doi: 10.1007/s001980050073. PMID 10024904